CLINICAL TRIAL: NCT05690295
Title: Comparison of the Effects of Prolonged Resistance-type Exercise Training Between Healthy Postmenopausal Women Versus Postmenopausal Women Survivors of Breast Cancer
Brief Title: Resistance-type Exercise Training in Postmenopausal Women Survivors of Breast Cancer
Acronym: MUSCLE-CLIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de La Frontera (Other)
Responsible Party: Principal Investigator, Gabriel Nasri Marzuca-Nassr, Professor, Universidad de La Frontera
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DFP22-0020
Record Dates: First submitted 2022-12-22; First posted 2023-01-19 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer Survivors; Postmenopause; Resistance Training
Keywords: breast cancer; hormone therapy; exercise; muscle mass; strength
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CLIMHEALTHY (Experimental): All postmenopausal women without breast cancer will be subjected to 12 weeks of full body resistance exercise training (3 times per week)
  Interventions: Other: Prolonged resistance-type exercise training
- CLIMCANCER (Experimental): All postmenopausal women survivors of breast cancer without or with Hormone Therapy (pecifically Aromatase Inhibitor or Tamoxifen) will be subjected to 12 weeks of full body resistance exercise training (3 times per week)
  Interventions: Other: Prolonged resistance-type exercise training

INTERVENTIONS:
Other: Prolonged resistance-type exercise training — All volunteers will be subjected to 12 weeks of whole-body resistance-type exercise training (3x/wk).

SUMMARY:
Background: In postmenopausal women, an alteration in body composition occurs as a consequence of the secretion of low levels of serum estrogens by the ovaries. Observing an increase in abdominal and mammary fat mass and a decrease in skeletal muscle mass, which is also accompanied by loss of muscle strength and physical function, which leads early to a sarcopenia.

On the other hand, the increase in estrogen production by adipose tissue has been associated with an increased risk of breast cancer during menopause because the mammary parenchyma is particularly sensitive to this type of estrogen. For this reason, Hormone Therapy (Aromatase Inhibitors and Tamoxifen) is prescribed in women with estrogen receptor-positive breast cancer. Antineoplastic treatments (Chemotherapy and Hormonal Therapy) have contributed to non-metastatic breast cancer currently presenting a high survival rate, not without adverse effects associated with the course of the disease, age and antineoplastic treatment, affecting various systems, but particularly skeletal muscle mass.

Therefore, resistance exercise training has been proposed as an effective intervention strategy to increase muscle mass and strength in different populations. However, the level of muscle response to this type of training in postmenopausal women survivors of breast cancer with and without hormone treatment (Aromatase Inhibitors and Tamoxifen) is unknown.

DETAILED DESCRIPTION:
Hypothesis: The increase in skeletal muscle mass after 12 weeks of progressive resistance-type exercise training is less in postmenopausal breast cancer survivors compared to healthy women of the same age range.

Postmenopausal breast cancer survivors without hormonal therapy will have greater gains in skeletal muscle mass compared to breast cancer survivors with Hormone Therapy (Aromatase Inhibitors or Tamoxifen) of the same age range after 12 weeks of progressive resistance-type exercise training.

Goals: The primary aim of this study is to compare the effects of a 12-week progressive resistance-type exercise training on muscle mass (whole body muscle mass) in healthy postmenopausal women versus postmenopausal women survivors of breast cancer with and without Hormone Therapy (Aromatase Inhibitors and Tamoxifen).

Specific goals Determine whether resistance-type exercise training can increase muscle strength and quality of life in healthy postmenopausal women versus postmenopausal women survivors of breast cancer with and without Hormone Therapy (Aromatase Inhibitors and Tamoxifen).

Identify whether circulating biochemical markers are up- or down-regulated in in healthy postmenopausal women versus postmenopausal women survivors of breast cancer with and without Hormone Therapy (Aromatase Inhibitors and Tamoxifen) after resistance-type exercise training

Methodology:

Study design Twenty-six postmenopausal women between 45 to 59 years will be divided into two groups: participants without cancer (CLIMHEALTHY, n=13) and participants survivors of breast cancer without or with Hormone Therapy (CLIMCANCER, n=13). All volunteers will be subjected to 12 weeks of whole-body resistance-type exercise training (3x/wk). Before, and after 12 weeks of training, whole-body dual energy x-ray absorptiometry (DEXA) scan will be performed for measured skeletal muscle mass and fasting blood samples will be obtained. Maximal strength will be determined by 1-repetition maximum (1RM), physical functioning by the short physical performance battery (SPPB) and quality of life by QLQ-BR23 at the same time points.

Study parameters/endpoints:

The main study endpoint is the increase in the skeletal muscle mass of whole-body assessed vial dual energy x-ray absorptiometry (DEXA).

Secondary endpoints include: Maximal strength assessment (1RM); Hand grip strength; Short physical performance battery (SPPB); quality of life (QLQ-BR23), Inflammatory and molecular markers (blood samples analysis).

Other study parameters include: Age, body weight, body height, body mass index (BMI), lipid profile, glucose, and insulin.

Expected results:

The impact of resistance-type exercise training to increase muscle mass in postmenopausal women survivors of breast cancer with or without hormonal therapy remains unclear. With the proposed project, the investigators expect that resistance-type exercise training will increase skeletal muscle mass, although the impact will be relatively lower in the participants survivors of breast cancer when compared with a group of healthy postmenopausal woman. The potential findings will define the efficacy of resistance-type exercise training to increase muscle mass in individuals with postmenopausal woman survivors of breast cancer. Better maintenance, or even an increase in muscle mass and strength increases independence, prolonging good health, recovery from disease and illness, and ultimately decreases burden on healthcare systems. These results will allow the creation of local, regional, national and international strategies to combat the adverse effects of breast cancer and its antineoplastic treatment, especially in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy postmenopausal women and postmenopausal women survivors of breast cancer with and without Hormonal Therapy (Aromatase Inhibitors and Tamoxifen) between 45 to 59 years.
* Women survivors of breast cancer with active Hormone Therapy in the last 12 months.
* Women breast cancer survivors with luminal molecular profile and positive estrogen receptors.
* Body mass index 18.5 < BMI < 30 kg/m2.
* Volunteers without cognitive impairment (abbreviated Minimental >13 points).

Exclusion Criteria:

* Active antineoplastic treatment in the last 12 months.
* >200 mL of volume difference between upper limbs and/or stage IV breast cancer.
* Performing regular resistance training (2 or more times per week, carrying out progressive training) in the previous 6 months.
* Cardiovascular diseases that are contradictory for physical activity (not included controlled Hypertension).
* All co-morbidities interacting with mobility and muscle metabolism of the body and that do not allow to (safely) perform the resistance-type exercise training (e.g. debilitating arthritis, spasticity/rigidity, all neurological disorders and paralysis).

Ages: 45 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 26 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
The changes in skeletal muscle thickness, including measurements for the biceps, triceps brachii, rectus femoris, vastus intermedius, and the total quadriceps, will be assessed using muscular ultrasound after prolonged resistance-type exercise training | Before, and after 12 weeks of training
  Measurements will be in centimeters.

SECONDARY OUTCOMES:
Change in kilograms of the arms strength measured via 1-Repetition Maximum (1RM) testing) after prolonged resistance-type exercise training | Before, and after 12 weeks of training
  Maximal strength assessment via 1RM testing of horizontal row, lat pull down and chest press exercises
Change in kilograms of the legs strength measured via 1-Repetition Maximum (1RM) testing) after prolonged resistance-type exercise training | Before, and after 12 weeks of training
  Maximal strength assessment via 1RM testing of leg press, and leg extension exercises
Change in kilograms of the hand grip strength measured via JAMAR handheld dynamometer after prolonged resistance-type exercise training | Before, and after 12 weeks of training
  Maximal strength assessment via 1RM testing of JAMAR handheld dynamometer
Change in points of the physical performance measured via Short physical performance battery (SPPB) after prolonged resistance-type exercise training | Before, and after 12 weeks of training
  Measurement of physical performance via SPPB, the minimum value is 0 point and the maximum value is 12 points. Higher score in the Physical Performance mean a better outcome and lower score mean a worse outcome
Change in points quality of life measured via questionnaire European Organisation for Research and Treatment of Cancer (EORTC QLQ-C30) after prolonged resistance-type exercise training | Before, and after 12 weeks of training
  Measurement of quality of life via EORTC QLQ-30, this questionnaire has 30 question covering functional state and cancer related symptoms. Besides, there are two specific question covering the "overall health" and "overall quality of life". The scores obtained are standardized and a score between 0 and 100 is obtained. High values on the global health and functional status scales indicate a better quality of life. However, high values on the symptom scale indicate a lower quality of life
Change in microgram per milliliter (µg/ml) of Human Insulin via ELISA after prolonged resistance-type exercise training | Before, and after 12 weeks of training
  Measurement in blood samples, the insulin will evaluate by ELISA using the Human Insulin ELISA Kit, following the manufacturer's recommendations
Change in milligrams per deciliter (mg/dL) of glucose via methods enzymatic-colorimetric | Before, and after 12 weeks of training
  Measurement in blood samples, the glucose will determined by enzymatic-colorimetric methods using an automatic photometer.
Change in milligrams per deciliter (mg/dL) of lipid profile via methods enzymatic-colorimetric | Before, and after 12 weeks of training
  Measurement in blood samples, the lipid profile will determined by enzymatic-colorimetric methods using an automatic photometer

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel N Marzuca-Nassr, Principal Investigator — Universidad de La Frontera
Locations (1):
- Department of Rehabilitation Sciences, Faculty of Medicine, Universidad de La Frontera. Temuco, Chile, Temuco, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Artigas-Arias M, Munoz-Cofre R, Vidal-Seguel N, Alegria-Molina A, Sapunar J, Curi R, Marzuca-Nassr GN. Resistance exercise training similarly improves work efficiency and measured submaximal oxygen consumption during the 6-min walk test in healthy postmenopausal women and breast cancer survivors. Eur J Appl Physiol. 2025 Sep 16. doi: 10.1007/s00421-025-05966-0. Online ahead of print. PMID 40954340
- [Derived] Artigas-Arias M, Alegria-Molina A, Vidal-Seguel N, Munoz-Cofre R, Carranza-Leiva J, Sepulveda-Lara A, Vitzel KF, Huard N, Sapunar J, Salazar LA, Curi R, Marzuca-Nassr GN. Skeletal muscle mass, strength, and physical performance gains are similar between healthy postmenopausal women and postmenopausal breast cancer survivors after 12 weeks of resistance exercise training. Support Care Cancer. 2024 Nov 23;32(12):818. doi: 10.1007/s00520-024-08973-7. PMID 39579274